CLINICAL TRIAL: NCT04489199
Title: Dijon Stroke Cohort
Acronym: DISCO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BEJOT 2020
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: CVA, Dijon Registry
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patient: Patient included in the Dijon Stroke Registry.
  Interventions: Other: Questionnaire and semi-structured interview

INTERVENTIONS:
Other: Questionnaire and semi-structured interview — questionnaire submitted by telephone 3 months, 6 months, 1 year, 5 years, and 10 years after the stroke/TIA. interview duration 20 to 40 minutes

SUMMARY:
The Dijon Stroke Registry, accredited by the Registry Evaluation Committee, INSERM and Public Health France, has been studying the epidemiology of cerebrovascular accidents (cerebral infarction, intracerebral haemorrhages, meningeal haemorrhages) and transient ischaemic attacks (TIAs) within the city of Dijon since 1985.

As a result of the development of therapies for acute disease, the prognosis of patients has improved over time. Thus, the number of stroke survivors has increased by 90% between the 1980s and today. This raises new issues: risk of vascular recurrence, drug iatrogeny, and functional impact of stroke for motor, cognitive or thymic function. In the absence of available data in France, the investigators wish to set up an extended cohort follow-up of patients in order to study their long-term prognosis and to study the impact of future therapies on the evolutionary course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* patients included in the Dijon Stroke Registry and not opposed to participating

Exclusion Criteria:

* minor patients; opposition to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the Dijon Stroke Registry
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Death rate | Trough study completion, an average of 10 years
Disability rate | Trough study completion, an average of 10 years
Quality of Life Questionnaire | Trough study completion, an average of 10 years
Neuropsychological questionnaire | Trough study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France